# "Optimization of Mass Drug Administration with existing drug regimens for Lymphatic Filariasis and Onchocerciasis"

## **Consent Script**

## 'DOLF' project, Death to Onchocerciasis and Lymphatic Filariasis

#### Sponsored by:

Bill and Melinda Gates Foundation: GH 5342

#### **Principal Investigator:**

Gary J. Weil, M.D.

**Version Number: 1.0** 

NCT Number: NCT01905436

Day Month Year: 23 Sep 2019

FOR IRB USE ONLY IRB ID #: 201107185 APPROVAL DATE: 09/23/19 RELEASED DATE: 09/23/19 EXPIRATION DATE: 09/21/20

## Questionnaire on resumption of mass treatment for parasitic infections in Foya district following the recent Ebola outbreak

**Invitation:** Because you are considered to be a leader in this community, you are being invited to participate in a survey to help understand the best way to resume mass treatment for parasitic infections following the recent Ebola epidemic. This program was started in 2012 to measure how these treatments improve the health of people in your village.

**Purpose**: The purpose of this questionnaire is to learn how your community feels about the mass treatment program that started in 2012 and their willingness to take the medicines when this public health program resumes in the near future. We would like to understand whether any actions or special education is needed to reassure your community about the purpose and value of this free drug distribution program. The project is being conducted by the Liberia Institute for Biomedical Research (LIBR) together with scientists at Washington University in Saint Louis, USA.

**Procedures**: During the questionnaire you will be asked questions about yourself, your community, mass drug administration programs, and Ebola. Your responses will be audio recorded. The questionnaire will take between 10-15 minutes. You may choose not to answer any question at any time. Your name will not be collected in the questionnaire.

**Risks**: There are no significant risks. Some of the questions may be uncomfortable or difficult for you to answer. You are not required to answer any question and may choose not to answer or stop the questionnaire at any time.

**Number of participants and duration of the project**: Approximately 100 adults will participate in the project. We will talk to 4 to 5 people per village in about twenty villages in Foya district over the course of 7 days.

**Benefits**: This information will benefit the Ministry of Health by providing information about how communities will respond to disease control programs that were interrupted by the Ebola epidemic. There is no direct benefit to you for participating in this survey. However by sharing your opinion you can help improve how mass drug administration programs operate in your community.

**Confidentiality**: Your name will not be recorded as part of the survey. Audio recordings and other information will be kept confidential and only made available to project researchers. Group results from this survey will be reported and (and perhaps published) without the names or identifying information of participants

**Participation is voluntary:** Your participation in this survey is entirely voluntary. Refusal to participate will not penalize you in any way, and you are free to withdraw at any time.

**Consent**: Your participation in this survey (answering our questions) will indicate that you have consented to join the survey.

Questions: You are free to ask any question regarding this questionnaire now. If questions arise later, please contact <u>Dr. Bolay</u>, who can be reached by telephone **Tel.** +2316516302 / +2316516803/ +231886513040 or Email: mailto: director.libr@gmail.com

**Note:** Program personnel must mark each computer record to verify that they have read this script to all participants and answered any questions. A copy of this information form should be left with each

FOR IRB USE ONLY IRB ID #: 201107185 APPROVAL DATE: 09/23/19 RELEASED DATE: 09/23/19 EXPIRATION DATE: 09/21/20

participant.